CLINICAL TRIAL: NCT04412187
Title: Inflammatory faCtors AfteR acUte Ischemic Stroke
Acronym: ICARUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Martin Dichgans (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital Muenster (Other)
Responsible Party: Sponsor-Investigator, Martin Dichgans, Prof. Dr. Martin Dichgans, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-428
Record Dates: First submitted 2020-05-22; First posted 2020-06-02 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Ischemic Stroke
Keywords: microglia; neuroinflammation; functional outcome after stroke
MeSH Terms: conditions — Ischemic Stroke; Neuroinflammatory Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 18 patients with cortical stroke and 18 patients with subcortical stroke
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TSPO PET imaging (Other): All study participants will receive [18F]-GE-180, i.e. TSPO PET imaging to assess microglia activation.
  Interventions: Diagnostic Test: [18F]-GE-180 PET; Diagnostic Test: 3T MRI; Diagnostic Test: immune cell profiling in blood

INTERVENTIONS:
Diagnostic Test: [18F]-GE-180 PET — serial [18F]-GE-180 PET imaging to assess microglia activation
  Other Names: TSPO PET imaging
Diagnostic Test: 3T MRI — serial MR imaging (i) to determine infarct characteristics, (ii) to identify gray and white matter structures connected to the infarct, (iii) to detect incident lesions, and (iv) to quantify longitudinal changes e.g. of cortical thickness
Diagnostic Test: immune cell profiling in blood — Cell-specific cytokine profiles, markers of activation, terminal differentiation as well as cytotoxicity will be assesses using flow cytometry.

SUMMARY:
ICARUS is an interventional single-centre hospital-based cohort study in patients admitted to the stroke unit with an acute ischemic stroke. The aims of the study are to i) define the characteristics and determinants of microglial activation after human stroke, and ii) assess the correlation of microglial activation with circulating inflammatory markers, structural brain changes on neuroimaging, and neurological outcomes.

ICARUS involves serial TSPO-PET imaging along with serial MRI, immune cell profiling in blood, and both clinical and laboratory assessments in 36 patients with acute ischemic stroke caused by a cortical (N=18) or strictly subcortical (N=18) infarct.

In a substudy, the investigators will include 10 independently recruited patients with acute ischemic stroke to assess MRI arterial spin labelling (ASL) sequences as a marker for perfusion measurement of the TSPO tracer.

DETAILED DESCRIPTION:
The neuroinflammatory response after ischemic brain injury has been identified as a pathomechanism in ischemic stroke. Stroke induces an activation of microglia in the brain, which lasts over months. However, the characteristics and mechanisms of this microglia activation are insufficiently defined.

Our study hypotheses are (i) that a subpopulation of patients with acute stroke develop prominent microglial activation, and (ii) that patients with extensive microglial activation are more likely to experience poor outcome.

Against this background, the investigators set up the "Inflammatory faCtors AfteR acUte ischemic Stroke (ICARUS)" study as an interventional single-centre hospital-based cohort study. N=36 patients with a cortical (N=18) or strictly subcortical (N=18) acute ischemic stroke will be recruited through the local stroke unit (Department of Neurology, LMU Munich). Study participation involves serial TSPO-PET imaging along with serial MR imaging, immune cell profiling in blood, and both clinical and laboratory assessments. Follow-up assessments at 3 weeks, 3 months, 6 months and 12 months will be conducted at the Institute for Stroke and Dementia Research (ISD) and at the Department of Nuclear medicine, both LMU Munich.

In a substudy, the investigators will include 10 independently recruited patients with acute ischemic stroke to assess MRI arterial spin labelling (ASL) sequences as a marker for perfusion measurement of the TSPO tracer. These patients will receive dynamic PET in addition to the ASL sequences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Acute ischemic stroke (time frame: <72 hours) as defined by an acute focal neurological deficit in combination with a corresponding infarct as documented by a diffusion weighted imaging (DWI)-positive lesion on magnetic resonance imaging (MRI); presence of an infarct involving the cortex or a strictly subcortical infarct
* Written informed consent prior to study participation
* Willingness to participate in study assessments including follow-up

Exclusion Criteria:

* Unwillingness or inability to give written consent
* Prior history of stroke, multiple infarcts, infratentorial infarcts affecting the brain stem or cerebellum
* Known diseases of the CNS other than stroke
* Immunomodulatory therapies within the last 3 months prior stroke
* Chronic inflammatory disease
* Infectious diseases within the last 7 days prior stroke
* Conditions interfering with follow-up such as end-stage malignancy
* Contraindications for MRI or PET (pacemaker, aneurysm clip, cochlear implant etc.)
* Radiation exposure of > 10mSv per year
* Pregnant or breastfeeding women
* Participation in a clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
microglia activation in patients with acute stroke | within 10 days after acute ischemic stroke
  Microglia activation will be assessed using TSPO PET imgaing.
microglia activation in patients with acute stroke | 3 months after acute ischemic stroke
  Microglia activation will be assessed using TSPO PET imgaing.
functional outcome in patients after acute ischemic stroke | 3 weeks after acute ischemic stroke
  Functional outcome measured by the modified Rankin Score (mRS) will be assessed and related to microglial activation.
functional outcome in patients after acute ischemic stroke | 3 months after acute ischemic stroke
  Functional outcome measured by the modified Rankin Score (mRS) will be assessed and related to microglial activation.
functional outcome in patients after acute ischemic stroke | 6 months after acute ischemic stroke
  Functional outcome measured by the modified Rankin Score (mRS) will be assessed and related to microglial activation.
functional outcome in patients after acute ischemic stroke | 12 months after acute ischemic stroke
  Functional outcome measured by the modified Rankin Score (mRS) will be assessed and related to microglial activation.
cognitive outcome in patients after acute ischemic stroke | 3 weeks after acute ischemic stroke
  Functional outcome in terms of cognition will be assessed by the Montreal Cognitive Assessment (MoCA) and related to microglial activation.
cognitive outcome in patients after acute ischemic stroke | 3 months after acute ischemic stroke
  Functional outcome in terms of cognition will be assessed by the Montreal Cognitive Assessment (MoCA) and related to microglial activation.
cognitive outcome in patients after acute ischemic stroke | 6 months after acute ischemic stroke
  Functional outcome in terms of cognition will be assessed by the Montreal Cognitive Assessment (MoCA) and related to microglial activation.
cognitive outcome in patients after acute ischemic stroke | 12 months after acute ischemic stroke
  Functional outcome in terms of cognition will be assessed by the Montreal Cognitive Assessment (MoCA) and related to microglial activation.

SECONDARY OUTCOMES:
inflammatory markers in blood | 3 weeks after acute ischemic stroke
  Inflammatory markers in blood will be assessed by flow cytometry and related to microglial activation.
inflammatory markers in blood | 3 months after acute ischemic stroke
  Inflammatory markers in blood will be assessed by flow cytometry and related to microglial activation.
Duplex ultrasound | 6 months after acute ischemic stroke
  Duplex ultrasound will be performed to assess potential progress of atherosclerosis related to inflammatory markers
3T MR imaging | 3 months after acute ischemic stroke
  3T MRI will be performed to relate infarct evolution, secondary neurodegeneration, and stroke outcome to microglial activation.
3T MR imaging | 12 months after acute ischemic stroke
  3T MRI will be performed to relate infarct evolution, secondary neurodegeneration, and stroke outcome to microglial activation.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Dichgans, Prof., Principal Investigator — LMU Munich; Peter Bartenstein, Prof., Principal Investigator — LMU Munich; Sibylle Ziegler, Prof., Principal Investigator — LMU Munich
Locations (2):
- Germany (2):
  - Insitute for Stroke and Dementia Research, Munich, Germany
  - Department of Nuclear Medicine, Munich

IPD SHARING:
Plan to Share IPD: Undecided